CLINICAL TRIAL: NCT03200015
Title: Effect of Metformin in Combination With R-CHOP for the First Line Treatment of Patients With Diffuse Large B-cell Lymphoma
Brief Title: Rituximab, Cyclophosphamide, Vincristine and Prednisone (R-CHOP) Plus Metformin in Diffuse Large-B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE16-00019
Record Dates: First submitted 2017-05-24; First posted 2017-06-27 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin arm (Experimental): Metformin 850 mg tablets. Initial dose 425 mg twice a day for 1 week, followed by 850 mg twice a day for 1 week, titrated to a maximum dose 850 mg every 8 hours until disease response evaluation study date (Computed tomography or positron emission tomography)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Potentially increasing the efficacy and safety of standard chemotherapy through several mechanisms

SUMMARY:
Evaluation of the safety and effectiveness of metformin as an adjunct to RCHOP chemotherapy for patients with newly diagnosed diffuse large-B cell lymphoma

DETAILED DESCRIPTION:
Patients with newly diagnosed diffuse large-B cell non Hodgkin lymphoma, irrespective of cell of origin status will receive metformin in combination to Rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone (RCHOP) chemotherapy for 6 cycles, until response evaluation as reported elsewhere:

1.- Rituximab 375 mg/m2 IV, day 1. 2.- Cyclophosphamide 750 mg/m2 IV, day 1. 3.- Doxorubicin 50 mg/m2 IV day 1. 4.- Vincristine 1.4 mg/m2 IV (2 mg maximum dose). 5.- Prednisone 60 mg/m2 PO days 1-5. Six cycles every 21 days.

Metformin will be added and administered in an outpatient basis, starting with 425 mg twice a day for 1 week, followed by 850 mg twice a day for 1 week, and lastly 850 mg every 8 hours maximum dose until re-staging. Laboratory tests will be performed serially.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed nodal diffuse large-B cell non Hodgkin lymphoma according to the 2008 World Health Organization classification for lymphoid malignancies
* No previous treatment other than prednisone or equivalent glucocorticoid up to 60 mg/m2 for 14 days
* Good performance status (Eastern Cooperative Oncology Group scale 0-2)
* Life expectancy >6 months
* Independently of the diagnosis of diabetes mellitus (any type)

Exclusion Criteria:

* History of intolerance or hypersensitivity reactions to metformin
* Primary central nervous system lymphoma
* History of other previous malignant neoplastic diseases <5 years prior to enrollment
* Evidence of systemic infection at the time of study
* HIV, hepatitis C or B virus infection
* Aspartate transaminase or alanine transaminase >2x upper limit of normal, bilirubin >2.5 times upper limit of normal
* Serum creatinine >1.5 mg/dL or chronic renal disease
* Cardiac insufficiency (New York Heart Association scale >1 or ejection fraction <50%)
* History of transformation from an indolent lymphoma
* Pregnancy
* History of lactic acidosis or alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2019-01-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Response rates | 6 months
  Overall, partial and complete responses to chemoimmunotherapy

SECONDARY OUTCOMES:
Progression-free survival | 2-5 years
  Survival with freedom from progression
Overall survival | 2-5 years
  Survival from diagnosis until death or last follow-up
Event-free survival | 2-5 years
  Survival from diagnosis until death or progression
Time to progression or relapse | 2-5 years
  Time from diagnosis until disease progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: David Gómez-Almaguer, MD, Study Chair — Hospital Universitario Dr. José Eleuterio González
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
No plans for a sharing plan pre-determined

REFERENCES:
- [Background] Asensio-Lopez MC, Lax A, Pascual-Figal DA, Valdes M, Sanchez-Mas J. Metformin protects against doxorubicin-induced cardiotoxicity: involvement of the adiponectin cardiac system. Free Radic Biol Med. 2011 Nov 15;51(10):1861-71. doi: 10.1016/j.freeradbiomed.2011.08.015. Epub 2011 Aug 25. PMID 21907790
- [Background] Shi WY, Xiao D, Wang L, Dong LH, Yan ZX, Shen ZX, Chen SJ, Chen Y, Zhao WL. Therapeutic metformin/AMPK activation blocked lymphoma cell growth via inhibition of mTOR pathway and induction of autophagy. Cell Death Dis. 2012 Mar 1;3(3):e275. doi: 10.1038/cddis.2012.13. PMID 22378068
- [Background] Alkhatib Y, Abdel Rahman Z, Kuriakose P. Clinical impact of metformin in diabetic diffuse large B-cell lymphoma patients: a case-control study. Leuk Lymphoma. 2017 May;58(5):1130-1134. doi: 10.1080/10428194.2016.1239822. Epub 2016 Oct 5. PMID 27701994
- See also: Similar study registered in Clinical trials.gov — https://clinicaltrials.gov/ct2/show/record/NCT02531308